CLINICAL TRIAL: NCT06608576
Title: Effects of Telematic Support in Physical Therapy Early Intervention on Infants At Risk of Neurodevelopmental Delays and Disorders
Brief Title: Telematic Support in Early Intervention on Infants At Risk of Neurodevelopmental Delays
Acronym: BBL-ATOP
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad de Granada (Other)
Collaborators: Hospital Universitario San Cecilio de Granada (Unknown)
Responsible Party: Principal Investigator, Marie Carmen Valenza, PT, PhD, Professor at University of Granada, Universidad de Granada
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: BBL-ATPO-2023
Record Dates: First submitted 2024-09-19; First posted 2024-09-23 (Actual); Last update posted 2024-09-23 (Actual); Status verified 2024-09

CONDITIONS: High-risk Infants
Keywords: early intervention; telerehabilitation; physical therapy; child development

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Standard Treatment (Active Comparator): participants will receive face-to-face early intervention treatment on physical therapy area once a month for two months.
  Interventions: Other: Face-to-face standard treatment
- Telematic Support (Experimental): Participants will receive weekly telematic early intervention sessions at home via video conferencing for two months.
  Interventions: Other: Telematic Support

INTERVENTIONS:
Other: Face-to-face standard treatment — Individualized early intervention treatment on physical therapy area as usual in the early intervention facilities once a month for two months. Instructions will be given to the parents for follow-up at home to stimulate the baby's motor development until next face-to-face session.
  Arms: Standard Treatment
Other: Telematic Support — The physiotherapist in charge of the telematic sessions will review and guide in real time through WhatsApp platform, the performance and active participation of the parents in the therapeutic activities being asked to follow-up at home in the face-to-face appointment, correcting, as necessary.
  Arms: Telematic Support

SUMMARY:
The purpose of this study is to evaluate the effects of early intervention support sessions via video conferencing as an adjuvant option to motor development on infants at risk of neurodevelopmental delays or disorders.

DETAILED DESCRIPTION:
The parents will be informed about the procedure and will be given a written informed consent in order to participate in the study. Then, the families will be randomized into one of two groups: standard treatment or telematic support. Both treatments in a 2-month period.

ELIGIBILITY:
Inclusion Criteria:

* Minor infants with a chronological or corrected age of 3 to 12 months and their parents attending physical therapy early intervention protocol at the Neuropediatrics and Neurodevelopment Unit of San Cecilio University Hospital in Granada.
* At risk of neurodevelopmental delays or disorders.
* Whose family has a cell phone with WhatsApp Application installed and internet to be able to carry out the telematic tests.

Exclusion Criteria:

* Independent walking children.
* Minor infants with diagnosis of neuromotor injury, visual and auditory sensory disorders or congenital anomalies.
* Infants with orthoses and/or prostheses.
* Children with health complications that enable the child's participation in the study.
* Not spanish-speaking parents.

Ages: 3 Months to 12 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Estimated)
Dates: Start 2024-02-15 (Actual); Primary Completion 2025-07-31 (Estimated); Study Completion 2025-07-31 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline in Motor Development on the Motor scale of the Infant Motor Development on the Bayley Scales of Infant and Toddler Development-III® (BSID-III) at month 2. | Baseline and Month 2.
  The BSID-III is an assessment tool for diagnosing developmental delays in early childhood from 1 to 42 months. It assesses 5 developmental domains: Cognitive Scale, Language Scale, Motor scale, Social-Emotional Scale and Adaptative Scale. The motor scale has 66 items in the fine motor and 72 items in the gross motor domain which are administrated according to the child development. Change= (2 months development score - baseline Score).
Change from Baseline in maturation of motor skills on the Alberta Infant Motor Scale (AIMS) at month 2. | Baseline and Month 2.
  The AIMS is an observational assessment tool that requires minimal handling of an infant by the examiner. It assesses the maturation of infant's motor skills from term (40 weeks gestation) to 18 months. It has 58 observational items divided into four subscales which are prone, supine, sitting and standing. Change= (2 months development score - baseline Score).
Change from Baseline in infant motor behaviour and motor development on the Infant Motor Profile (IMP) at month 2. | Baseline and Month 2.
  The IMP is a video-based assessment for infants aged 3 to 18 months. It assesses the spontaneous motor behaviour in supine, prone, sitting, standing, walking and during reaching and grasping - depending on the age of the infant. Includes 5 domains: the size of the infant's motor repertoire, the infant's ability to make an adaptive selection out of his/her repertoire, performance, symmetry and fluency. Change= (2 months IMP total and subscales scores - baseline scores).

SECONDARY OUTCOMES:
Change from Baseline in parents' quality of life on the Care-related quality of life (CarerQol) at month 2. | Baseline and Month 2.
  CarerQol measures the impact of providing informal care on caregivers. Consists of seven items questionnaire to evaluate the impact of informal care on satisfaction, support, problems with daily activities, and financial, relational, mental health and physical health problems of caregivers, and a Visual Analogue Scale which measures general well-being in terms of happiness from 0 (completely unhappy) to 10 (completely happy). Change= (2 months scores on each item - baseline Score).
Change from Baseline in levels of stress experienced by parents on the Parental Stress Scale (PSS) at month 2. | Baseline and Month 2.
  The Paretal Stress Scale is an 18-item self-report measure design to assess the perceived levels of stress resulting from being a parent. Overall possible scores on the scale range from 18 to 90 with higher scores indicating a higher level of stress. There are no average scores or "cut-off's" for this tool. Change= (2 months stress score - baseline score).
Parents satisfaction with the telematic support service measured with the Client Satisfaction Questionnaire (CSQ-8). | Month 2
  The Client Satisfaction Questionnaire is an 8-item measure of client or consumer satisfaction with health and human services including governmental and public benefit programs and services. Overall possible scores on the scale range from 8 to 32 with higher scores indicating a higher level of satisfaction with the given service. There are no average scores or "cut-off's" for this tool.
Change from Baseline in parental self-efficacy and satisfaction of being a parent on the Parenting Sense of Competence (PSOC) at month 2. | Baseline and Month 2.
  PSOC is a self-report measure that uses 17 questions to measure how capable a caregiver feels as a parent and how satisfied they are with being a parent. Possible scores range from 17 to 102 with higher scores indicating a higher parenting sense of competency. There are no average scores or "cut-off's" for this tool. Change= (2 months sense of competence score - baseline score).

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Universitario San Cecilio de Granada, Granada, Granada, Spain